CLINICAL TRIAL: NCT01626131
Title: Exercise: A Novel Treatment for Combat PTSD
Brief Title: Exercise: A Novel Treatment for Combat Post Traumatic Stress Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding agency, DoD, determined that the study could not meet its enrollment numbers by the end of the grant.
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTRuST-Exercise
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: combat disorders; exercise therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise treatment (Experimental): Aerobic and resistance training
  Interventions: Behavioral: exercise training
- Stretching treatment (Experimental)
  Interventions: Behavioral: Stretching training

INTERVENTIONS:
Behavioral: exercise training — Participants will engage in 3 aerobic and resistance exercise sessions (~60-75 min total per session) weekly for 8 consecutive weeks.
  Aerobic exercise will be performed for 30 minutes on a treadmill 3 times weekly. Before beginning, 10 min of stretches will be performed. Each exercise bout will begin and end with a 5-min warm-up and 5-min cool-down on the treadmill, not included in the prescribed exercise duration.
  Eight resistance exercises will be performed immediately following the aerobic exercise: lat pulldown, triceps pushdown, seated chest press, upright row, bicep curls, leg press, shoulder press, and abdominal crunches. Participants will perform two sets of 10 repetitions of each. A rest interval of 60 seconds will be taken between exercises. Research staff will initially assist the participants in choosing the proper resistance to use, and weight will be increased once 15 repetitions can be performed while maintaining proper form.
  Arms: Exercise treatment
Behavioral: Stretching training — Participants will engage in stretching sessions that will focus on whole-body flexibility. Participants will perform 3 sessions per week (~60 min) of 3 sets of 14 stretches focused on the muscle groups targeted by the exercise training (i.e., deltoids, pectorals, lats, forearms and biceps, triceps, quadriceps, hamstrings, and groins). Each stretch will be performed for 20 seconds and a rest interval of 60 seconds will be taken between each set.
  Arms: Stretching treatment

SUMMARY:
The primary objective of this pilot intervention study is to examine the efficacy of exercise for reducing the symptoms of posttraumatic stress disorder (PTSD) and other psychiatric and somatic symptoms. The sample will be composed of veterans aged 18-65 with combat-related PTSD (N = 40). Participants will be randomly assigned to one of two groups. Participants in the exercise training group (n = 20) will receive three 60-75 minute sessions per week of combination aerobic and resistance training for eight weeks. In the control stretching group, participants (n = 20) will receive training in whole-body flexibility three times per week for eight weeks. Secondary objectives include 1) determining feasibility of the intervention (as measured by the percentage of prescribed days of exercise completed by each participant, and percentage of time exercising completed at the prescribed intensity and duration); 2) determining the influence of exercise training on aerobic fitness and strength in the sample; and 3) determining whether psychiatric/somatic symptom improvements are associated with improvements in fitness and strength. Finally, exploratory objectives will include examining whether exercise training can improve early signs of heart disease, and whether certain biomarkers (using MRI and fMRI data and inflammatory markers) are associated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65yr
2. Diagnosis of PTSD
3. CAPS >30
4. Reported combat exposure per the Deployment Risk and Resilience Inventory (DRRI)
5. Sedentary lifestyle (planned activity for purpose of health < 2 days/wk)
6. Capability of giving informed consent

Exclusion Criteria:

1. Abuse of alcohol or drugs
2. Homelessness
3. Significant cognitive impairment (e.g., MMSE score of ≤ 26) that would hinder ability to understand the protocol
4. Signs or symptoms of cardiovascular, metabolic or pulmonary disease that would preclude participating in the exercise, including uncontrolled hypertension (> 159/99 mm Hg)
5. Usage of beta blockers, which could influence the heart rate response to exercise
6. Any physical or mental health condition that would contraindicate participation in the study (e.g., musculoskeletal, orthopedic, and/or neuromuscular disorders)
7. High suicidality
8. Below cutoff on either STAI (<30) or PCL-M (<40)
9. Pregnancy or plans to become pregnant in the next 4 months
10. Excessive levels of physical activity assessed via interview and pedometer recording
11. Current treatment for PTSD (drug or counseling) for a duration of less than eight weeks
12. Clinically judged to be unsuitable for participation by the research physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by a reduction in symptoms of posttraumatic stress disorder. | from pre- to post-treatment during 8-week intervention.
  Efficacy will be determined by a reduction in posttraumatic stress disorder symptoms as measured by the Clinician-Administered PTSD Scale-2 (CAPS-2).

SECONDARY OUTCOMES:
Feasibility as measured by adherence to the intervention. | during the 8-week intervention
  Feasibility will be determined by adherence to the intervention as measured by participation ≥ 2 times per week at the prescribed intensity for ≥ 80% of the exercise bouts.
Efficacy as measured by improvements in strength and fitness. | from pre- to post-treatment during 8-week intervention.
  Efficacy will be determined by improvements in strength and fitness. Fitness will be measured as graded maximal treadmill VO2max test performance.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D. Youngstedt, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- 921 Assembly Street, 3rd Floor, Public Health Research Center, University of South Carolina, Columbia, South Carolina, United States